CLINICAL TRIAL: NCT05541952
Title: BCG Re-vaccination for Primary Tuberculosis Prophylaxis in the Prison Population
Acronym: PPT-BCG
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: New evidence points to a new candidate vaccine, with a superior trial to BCG.
Sponsor: Federal University of Mato Grosso (Other)
Collaborators: Stanford University (Other); Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Roberto D Oliveira, Professor Research, Federal University of Mato Grosso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U1111-1236-5940; 07657119.8.0000.0021 (Other: CAAE CEP/UFMS)
Record Dates: First submitted 2022-07-25; First posted 2022-09-15 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Latent Tuberculosis
Keywords: Latent tuberculosis infection; Clinical trial; BCG re-vaccination; Interferon gamma
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will receive the 0.1 milliliter (mL) dose of BCG vaccine intradermally in the deltoid muscle region at the lower insertion level on the upper outer face of the right arm. When this recommendation can not be followed, the participant will be excluded from the study.
  Interventions: Biological: BCG
- Control (No Intervention): Participants assigned to the control arm will not receive any intervention and will be followed up with QFT and Genexpert for the detection of Mtb infection or diagnosis of tuberculosis.

INTERVENTIONS:
Biological: BCG — Revaccination with BCG, using the immunobiological used in the Brazilian public health network, strain Russia.
  Arms: Intervention

SUMMARY:
In the last decade, the incidence of tuberculosis (TB) has declined in much of the world, but has increased in Central and South America. Since 2000, the prison population in these localizations has grown by 206%, the highest increase in the world. In the same period, the reported cases of TB among the prison population (PP) increased by 269%. The extraordinarily high risk of acquiring TB within prisons creates a health and human rights crisis for PP that also undermines broader TB control efforts. Same studies identified an annual incidence of 26,000 per 100,000 for latent TB infection (through conversion of the tuberculin skin test) and of 4,000 per 100,000 for active TB among the PP in the state of Mato Grosso do Sul. In view of the combination of a high rate of infection and development of active disease and a short period of incarceration (on average 3 years), primary prophylaxis with BCG revaccination may be a cost-effective alternative associated with mass screening for control of the disease. Recently, in a phase 2 clinical trial, the BCG vaccine was shown to be 45% effective in preventing sustained IGRA conversion in adolescents in South Africa. With this study, the investigators aim to evaluate the effectiveness of BCG revaccination for primary TB prophylaxis in healthy individuals exposed to an environment of high disease transmission. This is an open-label, randomized phase IV clinical trial involving 760 individuals from three prisons in the state of Mato Grosso do Sul. Participants will be monitored for 26 months to calculate vaccination effectiveness to reduce latent tuberculosis infection as measured through sustained IGRA conversion. By carrying out this clinical trial, the researchers intend to obtain scientific evidence that can contribute to the tuberculosis control policy in Brazil.

DETAILED DESCRIPTION:
A randomized, open-label, phase IV clinical trial involving 760 prisoners to determine whether vaccination (or revaccination) with BCG reduces the incidence of latent tuberculosis infection (LTBI), as measured by the sustained conversion of the controlled release test of interferon gamma (IGRA) QuantiFERON TB Gold In Plus Qiagen (QFT).

Participants will be randomized into two groups: intervention to receive the BCG vaccine or control, which will not receive intervention, and followed for 24 months through scheduled quarterly visits to identify QFT conversion. Additional information on treatment for latent tuberculosis infection (LTBi) or TB will be obtained from government databases (Notification grievances Information system and Latent Tuberculosis Infection Information System). Blood samples will be collected before randomization and every 6 months until the 24th month of follow-up or at the time of early departure from the correctional unit. When necessary, sputum samples will be collected and x-rays will be performed to evaluate suspected tuberculosis.

760 adults inmates , serving time in a closed regime, will be involved in the study. The main exclusion criteria are the contraindication of BCG vaccination and a positive result for QFT or HIV. Participants will be randomized 1:1 resulting in approximately 360 people per group.

The research will be carried out in three prisons in the state of Mato Grosso do Sul, Brazil, Jair Ferreira de Carvalho Penal Establishment (EPJFC), Campo Grande Penal Institute (IPCG), both located in Campo Grande and Dourados State Penitentiary (PED), located in Dourados. Currently, approximately 6,300 adult males are held in these prisons, with an annual QFT conversion rate of 36% and an estimated TB incidence of 3.8% per year.

ELIGIBILITY:
Inclusion Criteria:

* No previous prison history.
* Be locked up for a maximum of 3 months.
* Have at least 24 months of unfulfilled penalty in a closed regime.
* No history or evidence of any clinically significant systemic disease, or any acute or chronic disease that may affect the safety, immunogenicity, or efficacy of the study vaccine.
* No history of treatment for active TB or latent Mtb infection.
* No history or evidence of active TB.
* No history of autoimmune disease or immunosuppression.
* No immunosuppressant medication in the last 30 days before intervention (D0) - with the exception of inhaled and topical corticosteroids.
* No lesions or any localized dermal changes at the insertion of the deltoid muscle.
* No history of allergic disease or reactions, including eczema, probably exacerbated by any component of the study vaccine.

Exclusion Criteria:

* QuantiFERON TB Plus Qiagen positive (Ag-Nil ≥0.20 IU / mL in both tubes).
* Reagent and / or undetermined result for HIV testing.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-17 (Estimated); Primary Completion 2020-08-17 (Estimated); Study Completion 2020-08-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of Latent Tuberculosis Infection (LTBI) | 6 months after the intervention.
  Defined as the number of cases of LTBI detected during follow-up.

SECONDARY OUTCOMES:
Percentage of sustained IGRA conversion | 2 months
  Defined as two tests with an Ag-Nil result ≥0.35 International Unit per milliliter (UI/ml) (in both tubes).
Incidence of active tuberculosis | Through study completion, an average of 24 months
  Diagnosis of pulmonary tuberculosis by chest X-ray, or sputum culture, or Genexpert.

CONTACTS AND LOCATIONS:
Overall Officials: Julio HR Croda, PhD, Principal Investigator — Federal University of Mato Grosso
Locations (1):
- Roberto Oliveira, Dourados, Mato Grosso do Sul, Brazil